CLINICAL TRIAL: NCT03027648
Title: Cohort Study of Levonorgestrel-releasing Intrauterine System for the Treatment of Symptomatic Adenomyosis
Brief Title: Levonorgestrel-releasing Intrauterine System for the Treatment of Symptomatic Adenomyosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Lei Li, Associate Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-OBGYN-2014
Record Dates: First submitted 2017-01-15; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Adenomyosis
Keywords: levonorgestrel-releasing intrauterine system; adenomyosis
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- patients with LNG-IUS (Other): Placement of levonorgestrel-releasing intrauterine system
  Interventions: Procedure: Placement of levonorgestrel-releasing intrauterine system

INTERVENTIONS:
Procedure: Placement of levonorgestrel-releasing intrauterine system — All the patients accepted treatment of levonorgestrel-releasing intrauterine system

SUMMARY:
Objective: To investigate the effects of levonorgestrel-releasing intrauterine system (LNG-IUS) for symptomatic adenomyosis.

Methods: From December, 2006 to December, 2014, symptomatic patients of adenomyosis diagnosed (with dysmenorrhea and/or menorrhea) by transvaginal ultrasound in outpatient or inpatient clinics of Peking Union Medical College Hospital were given the treatment of LNG-IUS. Before and after placement of LNG-IUS, during each following period, all the parameters were recorded prospectively, including carrying status of IUS, symptoms and scores of dysmenorrhea, menstruation scores, biochemical indicators, physical parameters, menstruation patterns and adverse effects.

Primary outcome measures: symptoms and scores of dysmenorrhea and menorrhea

Second outcome measures: carrying status of IUS

ELIGIBILITY:
Inclusion Criteria:

* Women with regular menses
* Adenomyosis diagnosed via transvaginal ultrasound
* With severe dysmenorrhea (VAS ≥ 7) and/or menorrhea (pictorial chart scores >100)
* Duration of placement > 12 months
* Size of uterus by physical examination less than uterus of 12-week pregnancy

Exclusion Criteria:

* Desire for pregnancy or lactation
* With diagnosis of malignancies or precancerous lesions
* Acceptance of laparotomy
* Contraindication of placing levonorgestrel-releasing intrauterine system

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1100 (Actual)
Dates: Start 2006-12; Primary Completion 2014-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
improvement of symptoms of adenomyosis assessed by change from baseline visual analogue scale at 5 years after placement of levonorgestrel-releasing intrauterine system | 5 years after placement of levonorgestrel-releasing intrauterine system
  visual analogue scale for pain

SECONDARY OUTCOMES:
unplanned taking-out rate in percent of levonorgestrel-releasing intrauterine system | 5 years after placement of levonorgestrel-releasing intrauterine system
spontaneously expulsion rate in percent of levonorgestrel-releasing intrauterine system | 5 years after placement of levonorgestrel-releasing intrauterine system
improvement of symptoms of adenomyosis assessed by verbal rating scales for pain | 5 years after placement of levonorgestrel-releasing intrauterine system
  verbal rating scales for pain
improvement of symptoms of adenomyosis assessed by hemoglobin for menorrhea | 5 years after placement of levonorgestrel-releasing intrauterine system
  hemoglobin for menorrhea
improvement of symptoms of adenomyosis assessed by pictorial chart scores for menorrhea | 5 years after placement of levonorgestrel-releasing intrauterine system
  visual analogue scale for pain

CONTACTS AND LOCATIONS:
Overall Officials: Leng Jinghua, MD, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with researchers via online database

REFERENCES:
- [Derived] Li L, Leng J, Jia S, Lang J. Treatment of symptomatic adenomyosis with the levonorgestrel-releasing intrauterine system. Int J Gynaecol Obstet. 2019 Sep;146(3):357-363. doi: 10.1002/ijgo.12887. Epub 2019 Jun 27. PMID 31194884